CLINICAL TRIAL: NCT05315921
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Single Ascending Doses of OsrhAAT in Healthy Volunteers
Brief Title: Study of OsrhAAT or Placebo in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthgen Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: HY1003-2021-P1
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-04

CONDITIONS: Emphysema Secondary to Congenital AATD
Keywords: OsrhAAT

STUDY DESIGN:
Intervention Model Description: This is a phase 1, single-center, placebo-controlled, double-blind, randomized study to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of OsrhAAT by a single ascending dose (SAD) design in healthy adults.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- OsrhAAT 1 mg/kg IV (Experimental)
  Interventions: Drug: OsrhAAT 1 mg/kg IV
- OsrhAAT 3 mg/kg IV (Experimental)
  Interventions: Drug: OsrhAAT 3 mg/kg IV
- OsrhAAT 10 mg/kg IV (Experimental)
  Interventions: Drug: OsrhAAT 10 mg/kg IV
- OsrhAAT 20 mg/kg IV (Experimental)
  Interventions: Drug: OsrhAAT 20 mg/kg IV
- OsrhAAT 40 mg/kg IV (Experimental)
  Interventions: Drug: OsrhAAT 40 mg/kg IV
- OsrhAAT 60 mg/kg IV (Experimental)
  Interventions: Drug: OsrhAAT 60 mg/kg IV

INTERVENTIONS:
Drug: OsrhAAT 1 mg/kg IV — Drug: OsrhAAT 1 mg/kg IV A single dose of OsrhAAT 1 mg/kg IV infusion at a rate approximately 0.04 ml/min/kg.
  Placebo: Normal Saline (0.9% Sodium Chloride)
  Arms: OsrhAAT 1 mg/kg IV
Drug: OsrhAAT 3 mg/kg IV — Drug: OsrhAAT 3 mg/kg IV A single dose of OsrhAAT 3 mg/kg IV infusion at a rate approximately 0.04 ml/min/kg.
  Placebo: Normal Saline (0.9% Sodium Chloride)
  Arms: OsrhAAT 3 mg/kg IV
Drug: OsrhAAT 10 mg/kg IV — Drug: : OsrhAAT 10 mg/kg IV A single dose of OsrhAAT 10 mg/kg IV infusion at a rate approximately 0.04 ml/min/kg.
  Placebo: Normal Saline (0.9% Sodium Chloride)
  Arms: OsrhAAT 10 mg/kg IV
Drug: OsrhAAT 20 mg/kg IV — Drug: OsrhAAT 20 mg/kg IV A single dose of OsrhAAT 20 mg/kg IV infusion at a rate approximately 0.04 ml/min/kg.
  Placebo: Normal Saline (0.9% Sodium Chloride)
  Arms: OsrhAAT 20 mg/kg IV
Drug: OsrhAAT 40 mg/kg IV — Drug: OsrhAAT 40 mg/kg IV A single dose of OsrhAAT 40 mg/kg IV infusion at a rate approximately 0.04 ml/min/kg.
  Placebo: Normal Saline (0.9% Sodium Chloride)
  Arms: OsrhAAT 40 mg/kg IV
Drug: OsrhAAT 60 mg/kg IV — Drug: OsrhAAT 60 mg/kg IV A single dose of OsrhAAT 60 mg/kg IV infusion at a rate approximately 0.04 ml/min/kg.
  Placebo: Normal Saline (0.9% Sodium Chloride)
  Arms: OsrhAAT 60 mg/kg IV

SUMMARY:
A Phase 1, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Single Ascending Doses of OsrhAAT in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be enrolled in the trial:

1. Able to understand and willing to sign the ICF
2. Healthy subjects, male or female, non-smokers, 18-55 years of age
3. No significant medical history, and in good health as determined by detailed medical history (neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease), full physical examination, vital signs, 12-lead electrocardiogram (ECG), urinalysis and laboratory tests at screening. For eligibility purposes, abnormal laboratory or vital signs results may be repeated once if abnormal result is observed at the initial reading. Moreover, abnormalities found in the ECG may need to be confirmed by repeated measurements.
4. Adequate organ function according to the following laboratory values:

   * Bone marrow function (absolute neutrophil count ≥1500/mm3 and platelet count ≥100,000/mm3).
   * Alanine aminotransferase (ALT) 7-56 units per liter of serum ( or institutional equivalent), AST 5-40 units per liter of serum (or institutional equivalent), alkaline phosphatase 20-140 units per liter of serum (or institutional equivalent), total bilirubin 0.1-1.0 mg/dL (or institutional equivalent) and creatinine clearance (Cockcroft-Gault equation) ≥90mL/min.
5. Female of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is 1 year of post-menopausal with a FSH > 40mIU/mL, or surgically sterile [defined as having a bilateral oophorectomy, hysterectomy or tubal ligation]) or agree to one of the following to prevent pregnancy and, if a woman of childbearing potential, have a negative pregnancy test at screening:

   * Practicing abstinence which is the preferred and usual lifestyle of the subject
   * If a sexually active woman of childbearing potential (sexually active with a non-sterile male partner) agrees to prevent pregnancy by using double methods of contraception as follow until 180 days after the administration of the investigational product:

     1. Simultaneous use of intra-uterine contraceptive device, placed at least 4 weeks prior to study drug administration, and condom for the male partner.
     2. Simultaneous use of hormonal contraceptives, starting at least 4 weeks prior to study drug administration and must agree to use the same hormonal contraceptive throughout the study, and condom for the male partner.
     3. Simultaneous use of diaphragm with intravaginally applied spermicide and male condom for the male partner, starting at least 21 days prior to study drug administration. Male subjects who are not vasectomized for at least 6 months and who are sexually active with a non-sterile female partner must agree to use double methods of contraception below from the first dose of randomized study drug until 120 days after their dose and must not donate sperm during their study participation period:

     <!-- -->

     1. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives (used since at least 4 weeks) or intra-uterine contraceptive device (placed since at least 4 weeks)
     2. Simultaneous use of a male condom and, for the female partner, a diaphragm with intravaginally applied spermicide
6. Body mass index (BMI) 18.0-32.0 kg/m2 and body weight ≥ 50.0 kg for males and

   * 45.0 kg for females
7. Blood pressure ≤ 139/89 mm Hg
8. Able to follow the study protocol and complete the trial

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be enrolled:

1. History of severe infection within 4 weeks prior to administration; signs and symptoms of any active infection regardless of severity within 2 weeks prior to administration.
2. History of hypersensitivity to OsrhAAT or any excipient or similar drugs
3. Known History of hypersensitivity to rice
4. Use of any prescription drugs, herbal supplements, or nonprescription drugs, including oral antihistamines (for seasonal allergies), within 1 month or 5 half-lives (whichever is longer) prior to study drug administration, or dietary supplements within 1 week prior to study drug administration, unless, in the opinion of the Investigator and the Sponsor, the medication will not interfere with the study. Over-the-counter multivitamins will be permitted. If needed, paracetamol/acetaminophen may be used, but must be documented in the Concomitant medications/Significant non-drug therapies page of the source data. Any questions of concomitant medications should be directed to the Sponsor.
5. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
6. Donation of blood 12 week prior to dosing
7. Pregnant, or nursing females
8. A history of psychiatric and psychological condition that, in the judgment of the Investigator, may interfere with the planned treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications
9. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms], Bazett Formula: QTc=QT/RR0.5）
10. Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer< 1000 cps/mL or 200 IU/mL), or cured Hepatitis C (negative HCV RNA test) may be enrolled, in the judgement of the Investigator.
11. Known infection with human immunodeficiency virus (HIV) and a cluster of differentiation 4 (CD4) count that is unknown or documented to be < 350 cells/mm3 within 12 months, or an Acquired Immune Deficiency Syndrome (AIDS)-defining illness
12. Known history of severe IgA deficiency
13. Immunization with a live or attenuated vaccine is prohibited within 4 weeks prior to study drug administration. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed
14. Receipt of an immunoglobulin or blood product 90 days prior to dosing
15. History of consuming more than 14 units of alcoholic beverages per week or of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits). Consumed > 3 (male) or 2 (female) units of alcohol as determined by blood alcohol testing at screening
16. History of significant drug abuse within one year prior to screening
17. Positive urine drug screen (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, cotinine and opiates)
18. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence of adverse events (AEs), serious adverse events (SAEs), and infusion site reactions | Adverse events (AE) will be collected from the time of informed consent until EOS. SAE will be collected by the Investigator from the informed consent through 180 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No